CLINICAL TRIAL: NCT05277740
Title: Implementation of a Novel Functional Eye-Tracking Biomarker for Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Innodem Neurosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-7045; ETNA-CIS (Other: McGill University)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Clinically Isolated Syndrome; Relapsing Remitting Multiple Sclerosis
Keywords: multiple sclerosis; clinically isolated syndrome; eye-tracking
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CIS: Diagnosis of Clinically Isolated Syndrome (CIS) with abnormal MRI.
  Interventions: Device: Eye-tracking
- RRMS: Diagnosis of Relapsing-Remitting MS (RRMS).
  Interventions: Device: Eye-tracking
- Healthy Control: Participant with no evidence or history of significant neurodegenerative disorder affecting brain function.
  Interventions: Device: Eye-tracking

INTERVENTIONS:
Device: Eye-tracking — Eye-tracking technology and algorithms used to successfully capture and track eye movements using an electronic tablet and the embedded camera of the device.

SUMMARY:
This study aims to develop and validate a sensitive and non-invasive eye-tracking software application.

This study will obtain participant responses to brief cognitive tests designed to evaluate several key functions known to be affected by CIS and RRMS and non-invasive eye movement measurements in response to visually presented stimuli during specifically designed eye-tracking tests. The study data will be used to develop machine learning algorithms and validate a software application intended to identify which metrics-or combination thereof-can serve as reliable biomarker of CIS and RRMS disease progression and cognitive status.

ELIGIBILITY:
Inclusion Criteria:

* For all participants

  1. Able to provide informed consent
  2. Visual acuity of 20/100 in at least one eye (corrective glasses, contact lenses, surgery etc. are permitted)
* For patients only

  1. Confirmed diagnosis of CIS with abnormal MRI or RRMS
  2. Neurological condition is medically stable during the study visit

Exclusion Criteria:

* For all participants:

  1. Evidence or medical history of psychiatric issues, which are known to also affect movements and oculomotor control.
  2. Aged above 65 or less than 18 years of age.
  3. Presence of comorbid neurological conditions to avoid eye movement anomaly confounds (Strabismus, cranial nerve palsy, stroke-causing hemianopsia).
  4. Diagnosis of macular edema or other pre-existing ocular conditions that would prevent from performing the eye movement assessments.
* For healthy controls only:

  1. Evidence or history of significant neurological disorder (Multiple Sclerosis, Parkinson's Disease, Amyotrophic Lateral Sclerosis, Dementia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target sample size for the CIS group is 45. The target sample size for the RRMS group is 45. Data will also be acquired from a control group (n=30) that will be frequency-matched for age.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Symbol Digit Modalities Test (SDMT) score at Month 12 | Baseline and Month 12
  The SDMT is used to assess divided attention, visual scanning, tracking and motor speed. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Scoring involves summing the number of correct substitutions within the 90 second interval.
  The SDMT is used to assess divided attention, visual scanning, tracking and motor speed. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Scoring involves summing the number of correct substitutions within the 90 second interval.
  The SDMT is used to assess divided attention, visual scanning, tracking and motor speed. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Scoring involves summing the number of correct substitutions within the 90 second interval.

SECONDARY OUTCOMES:
Change from Baseline in the Expanded Disability Status Scale (EDSS) score at Month 12 | Baseline and Month 12
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Change from Baseline in the Brief International Cognitive Assessment for MS (BICAMS) scores at Month 12 | Baseline and Month 12
  The BICAMS is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment. It includes the Symbol Digit Modalities Test (SDMT), the California Verbal Learning Test-2 (CVLT2) and the Brief Visuospatial Memory Test-Revised (BVMT-R)
Change from Baseline in the Multiple sclerosis functional composite (MSFC) scores at Month 12 | Baseline and Month 12
  A clinical trial outcome measure of assessing the severity of multiple sclerosis (MS) primarily. used in research. The score is based on a combination of timed tests of walking, arm function, and cognitive ability. It is a three-part, standardized, quantitative, assessment instrument for use in clinical studies, particularly clinical trials, of MS. The MSFC can produce scores for each of the three individual measures as well as a composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Giacomini, MD, Principal Investigator — McGill University
Locations (1):
- Montreal Neurological Institute and Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified metrics (e.g. age, medication intake, cognitive scores) will be uploaded onto a secure could-based server of collaborator (Innodem) for data analysis purposes, and will not be shared with anyone other than the collaborator.